CLINICAL TRIAL: NCT00430833
Title: Candesartan Use in Hypertrophic and Non-Obstructive Cardiomyopathy Estate (The CHANCE): a Double-Blind, Placebo-Controlled, Randomized, Multicenter Study
Brief Title: CHANCE - Candesartan in Hypertrophic Cardiomyopathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charles University, Czech Republic (Other)
Collaborators: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 9164
Record Dates: First submitted 2007-01-31; First posted 2007-02-02 (Estimated); Last update posted 2007-02-02 (Estimated); Status verified 2007-01

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — candesartan

INTERVENTIONS:
Drug: candesartan

SUMMARY:
The primary hypothesis of the study is that treatment with AT1-R antagonist in patients with nonobstructive form of HCM will be first save, second will cause regression of myocardial hypertrophy.

DETAILED DESCRIPTION:
Patients will be randomly assigned in 1:1 ratio either to candesartan (target dose 32 mg once daily) or matching placebo. The initial dose of the study drug will be 8 mg once daily. Study drug dose will be then doubled as tolerated every 2 weeks while aiming for a target dose of 32 mg once daily. Monitoring of blood pressure, serum creatinine, serum potassium and pressure gradient in LV outflow tract will be performed during dose increase. Patients will be observed clinically at 3, 6, and 12 months after the maintenance dose was reached. Exercise tolerance will be assessed by bicycle ergometry, presence of malignant arrhythmias by Holter monitoring, extent of LV hypertrophy by 2-dimensional echocardiography, and LV outflow tract pressure gradient by Doppler echocardiography at baseline and 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* HCM defined on the basis of echocardiographic criteria showing a nondilated, hypertrophied left ventricle (any wall thickness > 15 mm) in the absence of known causes of LV hypertrophy hypertension or valvular disease

Exclusion Criteria:

* Hypertrophic obstructive cardiomyopathy defined as presence of resting gradient in left ventricular outflow tract ³30 mmHg or in righ ventricular outflow tract ³15 mmHg at Doppler echocardiography;
* Atrial fibrillation;
* Treatment with ACE inhibitors or AT1-R antagonists any time in the past;
* Contraindications to AT1-R antagonists;
* Coronary artery disease, renal failure, hepatic disorders or serious intercurrent illness limiting survival; and
* Poor echocardiographic image quality.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Martin Penicka, PhD, Principal Investigator — Charles University, Prague, Czech Republic
Locations (1):
- Cardiocenter, Third Faculty of Medicine, Charles University, Prague, Czechia

REFERENCES:
- [Derived] Penicka M, Gregor P, Kerekes R, Marek D, Curila K, Krupicka J; Candesartan use in Hypertrophic And Non-obstructive Cardiomyopathy Estate (CHANCE) Study Investigators. The effects of candesartan on left ventricular hypertrophy and function in nonobstructive hypertrophic cardiomyopathy: a pilot, randomized study. J Mol Diagn. 2009 Jan;11(1):35-41. doi: 10.2353/jmoldx.2009.080082. Epub 2008 Dec 12. PMID 19074594